CLINICAL TRIAL: NCT01058265
Title: Effect of an Integrative Medicine Consultation on Outcome for Patients With Pain or Fatigue
Brief Title: Integrative Medicine Consultation for Patients With Pain or Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Larry Bergstrom, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-008497
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-01

CONDITIONS: Pain; Fatigue
MeSH Terms: conditions — Pain; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrative (Experimental): Integrative Medical care is defined as a comprehensive medical evaluation that emphasizes wellness and healing of the whole person as major goals above and beyond suppression of a specific somatic disease. The patient is viewed as a whole person with mind and spirit as well as body and these dimensions are incorporated into diagnosis and treatment plans. An integrative medicine evaluation includes four aspects of health: physical, emotional, mental and spiritual health. Maximum improvement in health is achieved by addressing each aspect through an integrated treatment plan. The evaluation generally takes 90-120 minutes.
  Interventions: Other: Integrative
- Standard (Active Comparator): Standard general medical evaluation.
  Interventions: Other: Standard

INTERVENTIONS:
Other: Integrative — Integrative Medicine medical evaluation.
  Arms: Integrative
Other: Standard — Standard general medical evaluation.
  Arms: Standard

SUMMARY:
Patients with a diagnosis of chronic fatigue or pain benefit minimally from a conventional medical evaluation yet consume a large amount of medical resources and time. The question is to see if patients with a diagnosis of chronic pain or fatigue benefit from an Integrative Medicine medical evaluation conducted by physician who has additional training in Integrative Medicine. Patients who call for a general medical examination with a complaint of chronic fatigue or pain will be set up with the integrative medical specialist or standard general medical evaluation.

ELIGIBILITY:
* Patients seeking a medical evaluation for a primary complaint of pain or fatigue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Bergstrom, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integrative | Standard
Started | 22 | 25
Completed | 11 | 13
Not Completed | 11 | 12
Not completed — Lost to Follow-up | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrative | Standard | Total
Number analyzed (Participants) | 22 | 25 | 47
Age Continuous [Median (Inter-Quartile Range); unit: Year] | 43.4 [28.8 to 53.3] | 51.8 [37.0 to 62.4] | 44.7 [34.8 to 57.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 20 | 22 | 42
  American Indian or Alaska Native | 0 | 1 | 1
  Other/Unknown | 2 | 2 | 4
Reason for appointment [Number; unit: Participants]
  Fatigue | 15 | 8 | 23
  Pain | 6 | 14 | 20
  Both | 1 | 3 | 4
Weight [Mean (Standard Deviation); unit: kg] | 70.5 (17.8) | 76.1 (24.6) | 73.6 (21.7)
Height [Mean (Standard Deviation); unit: cm] | 168.4 (8.1) | 161.3 (20.3) | 164.6 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: Short Form 36 (SF-36) Physical Component Summary (PCS)
Description: It yields an eight-scale profile of scores (physical functioning, social functioning, role-physical, role-emotional, bodily pain, general health, mental health, and vitality) as well as summary physical and mental measures (Ware et al., 1998). The Physical Component Summary ranges from 0 to 100, and higher score indicates better physical condition. It is based on norm-based scoring, which applies a transformation with mean equals to 50 and standard deviation equals to 10, and makes it possible to comparison.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Integrative | Standard
Number analyzed (Participants) | 11 | 13
Scores on a scale | 36.2 [22.2 to 44.1] | 39.0 [32.2 to 43.3]
Statistical Analysis 1: Comparison: Integrative vs Standard; The null hypothesis is that there is no difference in PCS between two groups; Test type: Superiority or Other; p = 0.487, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Short Form 36 (SF-36) Mental Component Summary (MCS)
Description: It yields an eight-scale profile of scores (physical functioning, social functioning, role-physical, role-emotional, bodily pain, general health, mental health, and vitality) as well as summary physical and mental measures (Ware et al., 1998). The Mental Component Summary ranges from 0 to 100, and higher score indicates better mental health status. It is based on norm-based scoring, which applies a transformation with mean equals to 50 and standard deviation equals to 10, and makes it possible to comparison.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Integrative | Standard
Number analyzed (Participants) | 11 | 13
Scores on a scale | 45.2 [36.4 to 50.8] | 47.9 [35.2 to 57.3]
Statistical Analysis 1: Comparison: Integrative vs Standard; The null hypothesis is that there is no difference in MCS between two groups; Test type: Superiority or Other; p = 0.817, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Three months
Description: Due to the nature of the study, the potential risk to the participants is minimal.
Arm/Group | Integrative | Standard
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/22 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes